CLINICAL TRIAL: NCT06509724
Title: Postoperative Conventional Versus Hypofractionated Intensity-modulated Radiation Therapy With Concurrent Chemotherapy in Cervical Cancer: A Prospective Multicenter Randomized Phase III Trial (POHIM_P3 Trial)
Brief Title: Comparison of Conventional and Hypofractionated IMRT in High-Risk Cervical Cancer Post-Radical Hysterectomy
Acronym: POHIM-P3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2024-04-058; KROG 24-05 (Other Grant/Funding Number: Korea Radiation Oncology Group)
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Fractionation Group (Active Comparator): The conventional fractionation group will receive 1.8-2.0G per session for a total of 25-28 sessions, amounting to 40-50.4Gy of radiation therapy. Chemotherapy will be administered once a week for a total of 5-6 sessions.
  This group are allowed to receive brachytherapy.
  Interventions: Radiation: Conventional Fractionated IMRT
- Hypofractionation Group (Experimental): The hypofractionation group will receive 2.5Gy per session for a total of 16 sessions, amounting to 40 Gy of radiation therapy. Chemotherapy will be administered once a week for a total of 3 sessions.
  This group are allowed to receive brachytherapy.
  Interventions: Radiation: Hypofractionated IMRT

INTERVENTIONS:
Radiation: Conventional Fractionated IMRT — * Dose: 1.8-2.0 Gy per session, total 25-28 sessions (40-50.4Gy)
  * Chemotherapy: Weekly, total 5-6 sessions
  Arms: Conventional Fractionation Group
Radiation: Hypofractionated IMRT — * Dose: 2.5 Gy per session, total 16 sessions (40Gy)
  * Chemotherapy: Weekly, total 3 sessions
  Arms: Hypofractionation Group

SUMMARY:
Radical hysterectomy and radiation therapy are standard treatments for cervical cancer. However, there are no reported studies on the frequency of side effects and treatment outcomes when hypofractionated radiation therapy and intensity modulated radiation therapy(IMRT) are used during radiation therapy.

Hypofractionated radiation therapy increases the daily dose and reduces the number of treatment sessions, which may increase the risk of side effects, but its safety has been confirmed in some cases of early cervical cancer and endometrial cancer. Additionally, applying IMRT, a technique designed to protect normal tissue, during concurrent chemoradiotherapy has shown positive results in reducing the incidence of acute side effects.

Investigators previously demonstrated that combining hypofractionated IMRT with chemotherapy for high-risk postoperative cervical cancer patients resulted in high survival rates and low toxicity in a phase 2 exploratory study. Base on this result, this study aimed to compare the efficacy and safety of conventional fractionated radiation therapy and hypofractionated radiation therapy.

DETAILED DESCRIPTION:
* This phase 3 multicenter randomized controlled trial evaluates two radiation therapy regiments in high-risk cervical cancer patients who have undergone radical hysterectomy. Participants are randomly assigned in a 1:1 ratio to receive either conventional fractionated IMRT(Intensity modulated radiation therapy) or hypo fractionated IMRT, both in combination with concurrent chemotherapy.
* The conventional fractionation group receives 1.8-2.0 Gy per session for a total of 25-28 sessions (total 40-50.4 Gy) with weekly chemotherapy (total 5-6 sessions). The hypofractionation group receives 2.5 Gy per session for a total of 16 sessions (total 40 Gy) with weekly chemotherapy (total 3 sessions). Brachytherapy is allowed in both group.
* Stratification factors for randomization include lymph node metastasis status and adenocarcinoma vs. non-adenocarcinoma. Blocked randomization will be used. The study aims to assess local control rates, overall, survival, disease-free survival, and acute and late toxicity profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed histologically with cervical cancer
* Patients diagnosed histologically with Squamous cell carcinoma, Adenocarcinoma, or Adenosquamous carcinoma
* Patients who have undergone radical hysterectomy and pelvic lymphadenectomy
* Patients who meet the indication for radiotherapy in postoperative pathological examination (at least on of the following):

A. Pelvic lymph node metastasis B. Parametrial involvement C. Positive surgical margins

* Adult aged 20 to 75 years
* Patients with an ECOG 0-1 within 1 week prior to study participation
* Maintained bone marrow function: granulocyte ≥1.0 x 103/µl, platelets ≥30 x 103/µl, hemoglobin ≥9.5 g/dl
* Maintained renal and liver function (Creatinine <2.0 mg/dL, Bilirubin < 1.5 mg/dl)
* Patients who have voluntarily signed the consent form

Exclusion Criteria:

* Patients with distance metastasis (including ovarian and para-aortic lymph node metastasis)
* Patients who have previously received radiotherapy to the pelvic area
* Patients who have undergone radical hysterectomy more than 3 months prior
* Patients with untreated serious acute illnesses (e.g., stroke, cerebral infarction, myocardial infarction) other than cervical cancer
* Patients who received neoadjuvant chemotherapy before surgery
* Patients who will not receive concurrent chemotherapy during radiotherapy
* Patients with a history of another cancer diagnosis within the past 5 years, except for thyroid cancer, skin cancer, or carcinoma in suit

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Local control rate for the radiation treatment area | Up to 3 years
  The percentage of patients who achieve local control of their cervical cancer within the radiation treatment area. Local control is defined as the absence of tumor recurrence or progression in the region.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  The duration of time from the date of randomization until death from any cause. This measure will evaluate the effectiveness of the treatment in prolonging life.
Disease-free survival (DFS) | Up to 5 years
  The length of time from the date of randomization until the occurrence of any signs or symptoms of cervical cancer, such as local recurrence, distant metastasis, or secondary cancer. This measure assesses the efficacy of the treatment in preventing cancer recurrence.
Acute Toxicity Profile | During treatment and up to 3 months post-treatment
  The incidence and severity of acute treatment-related toxicities, as measured by the Common Terminology Criteria for Adverse Events (CTCAE). Acute toxicities are those occurring within 90days of the start of treatment.
Late Toxicity Profile | From 3 months post-treatment up to 5 years
  The incidence and severity of late treatment-related toxicities, as measured by the Common Terminology Criteria for Adverse Events (CTCAE). Late toxicities are those occurring more than 90 days after the completion of treatment.
Quality of life (QoL) | Baseline, end of treatment, 6 months post-treatment, and annually up to 5 years
  Assessment of the patients' quality of life using validated questionnaires such as the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This measure evaluates the impact of treatment on the patients' overall well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

REFERENCES:
- [Derived] Cho WK, Park W, Lee JH, Kang HC, Yoon M, Eom KY, Kim YS, Park S, Kim YS, Kim YJ, Choi E, Kim DY. Postoperative conventional versus hypofractionated intensity-modulated radiation therapy with concurrent chemotherapy in cervical cancer: a prospective multicenter randomized phase III trial (POHIM_P3 trial). J Gynecol Oncol. 2026 Jan;37(1):e4. doi: 10.3802/jgo.2026.37.e4. Epub 2025 Jul 4. PMID 40676909